CLINICAL TRIAL: NCT00842309
Title: A Randomized, Double-blind, Placebo-controlled Trial of D-cycloserine Augmentation of Behavior Therapy for Body Dysmorphic Disorder
Brief Title: D-Cycloserine Augmentation of Behavior Therapy for Individuals With Body Dysmorphic Disorder
Acronym: BDD/DCS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008P001429
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Body Dysmorphic Disorder
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Active Comparator): 100mg of d-cycloserine in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  Interventions: Drug: d-cycloserine
- Placebo (Placebo Comparator): Placebo in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: d-cycloserine — 100mg of d-cycloserine in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  Other Names: seromycin
  Arms: D-cycloserine
Drug: Placebo — Placebo in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to conduct a double-blind, placebo-controlled study of D-cycloserine (DCS) augmentation of behavior therapy in individuals with Body Dysmorphic Disorder (BDD). Specifically, we intend to randomize 50 individuals with BDD to receive either DCS (n = 25) or placebo (n = 25) one hour prior to 8 of 10 behavior therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Primary diagnosis of Body Dysmorphic Disorder as determined by DSM-IV criteria
* BDD Yale-Brown Obsessive Compulsive Scale score greater than or equal to 24
* Females of childbearing potential must have a negative urinary beta-HCG test
* Subjects currently taking psychotropic medication must be on a stable does for at least two months prior to initiating study procedures

Exclusion Criteria:

* Pregnant or breastfeeding women will be excluded
* People taking medications that may interfere with DCS
* History of seizure disorder or other serious medical illnesses such as cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* Comorbid psychiatric diagnoses (alcohol dependence, bipolar disorder, psychosis, borderline personality disorder, organic mental disorder, or development disorder). If subjects have any other comorbid disorder, the BDD symptoms have to be the primary concern.
* Persons taking medications that may lower seizure threshold, including clozapine, pethidine, and the following antibiotics in high dosage: penicillins, cephalosporins, amphotericin, and imipenem
* Those deemed to pose a serious suicidal or homicidal threat will be excluded
* Current psychotherapy or failure to benefit from ten or more sessions of previous ERP treatment is a rule-out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-11; Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Mass General Hospital BDD clinic website — http://mghocd.org/
- See also: OCD and Related Disorders Clinic at MGH — http://www.mghocd.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants consented and screened. Of those, 28 were deemed eligible to participate and randomized to a condition. The remaining 40 participants were excluded for the following reasons: Did not meet criteria (n= 30) Declined to participate (n= 4) Did not show (n= 3) Other (n= 3)
Groups:
- D-cycloserine-augmented CBT: 100mg of d-cycloserine in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  d-cycloserine: 100mg of d-cycloserine in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
- Placebo-augmented CBT: Placebo in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
  Placebo: Placebo in pill form administered 1 hour before behavior therapy sessions once a week for 8 weeks.
Period: Overall Study
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Started | 14 (14 randomized. 2 withdrew prior to initiating DCS-not included in modified intent-to-treat analyses.) | 14
Completed | 11 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants included in modified intent-to-treat (ITT) analyses were 26 adults who completed at least one treatment session in their randomized condition [CBT plus DCS (n = 12); CBT plus placebo (n = 14)]. Note that 2 participants in CBT plus DCS did not complete any sessions in their randomized condition and were excluded from analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.92 (5.74) | 29.07 (11.04) | 26.69 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
BDD-YBOCS [Mean (Standard Deviation); unit: units on a scale] — The BDD-YBOCS is the gold-standard, semi-structured clinician-administered assessment of BDD severity. It contains 12 items ranging from 0 to 4, which are summed to generate a total score (range = 0 to 48). Higher scores indicate more severe BDD symptoms. The BDD-YBOCS will be used to assess change in BDD symptoms from baseline to endpoint.
  units on a scale | 31.75 (5.03) | 30.36 (4.45) | 31 (4.68)

OUTCOME MEASURES:

1. Primary Outcome: Body Dysmorphic Disorder Yale-Brown Obsessive Compulsive Scale (BDD-YBOCS)
Description: The BDD-YBOCS is the gold-standard, semi-structured clinician-administered assessment of BDD severity. It contains 12 items ranging from 0 to 4, which are summed to generate a total score (range = 0 to 48). Higher scores indicate more severe BDD symptoms. The BDD-YBOCS will be used to assess BDD symptoms at baseline and endpoint.
Time Frame: Endpoint (post-treatment, week 11)
Population: BDD-YBOCS was a clinician-administered measure administered to patients with body dysmorphic disorder.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 11 | 13
units on a scale | 19.64 (6.8) | 18.77 (10.03)

2. Primary Outcome: Body Dysmorphic Disorder Yale-Brown Obsessive Compulsive Scale (BDD-YBOCS)
Description: as for outcome 1
Time Frame: Mid-treatment (week 6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 12 | 13
units on a scale | 21.75 (5.34) | 20.85 (8.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at pretreatment, mid-treatment, post-treatment and at 1- and 6- month follow-up visits.
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine-augmented CBT (N=14) | Placebo-augmented CBT (N=14)
Feeling drowsy or sleepy (Nervous system disorders) | 0 (0) | 2 (2)
Depressive symptoms (Psychiatric disorders) | 1 (1) | 1 (1) — One patient experienced a major depressive episode during the follow-up period. Another patient had an increase in depressive symptoms and suicidal thoughts (no plan) during follow-up.
Stress fracture in both arms (General disorders) | 1 (1) | 0 (0)
Tendonitis in knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Went to dermatologist for acne and started medication (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT00842309/Prot_SAP_002.pdf